CLINICAL TRIAL: NCT00282958
Title: The Therapeutic Use of Botulinum Toxin Type A in Subacute Cervical/Upper Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAT0014
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Subacute Cervical Pain; Subacute Upper Back Pain
MeSH Terms: interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin type a (Botox)

SUMMARY:
To determine the therapeutic efficacy of Botox not only for chronic cervical/upper back pain but also for subacute pain.

DETAILED DESCRIPTION:
Subjects diagnosed with subacute (2-6 months post-onset) bilateral cervical/ upper back pain will be recruited in this double-blind control study.

A total of 30 subjects with subacute cervical/upper back pain will be recruited. If patients are qualified as participants and agreed to participate in the study by signing the consent form, they will be randomized into either (A) control group (injection of normal saline injection) or (B) study group (injection of BOTOX). The initial history taking step will include medical history including medication and surgery history, duration of pain, pre-injection neck disability index (NDI) and visual analogue scale (VAS) for pain. VAS score will be collected for 4 weeks before injection to ensure stable VAS, otherwise medical records will be reviewed to ensure stable feature of pain. Short Form (SF) -36 Health Survey will be used to assess functional status, and the Beck Depression Inventory (BDI) will be applied to assess psychological aspect. Physical examination will be performed to determine the most tender cervical/ upper back muscles, and rule out operative condition. A simple swallowing test (3-oz water swallowing test) will be applied for dysphagia screening.

The patients will be maintained with routine, standardized physical therapy, oral medication, and stretch exercise after the injection. NDI, VAS, and SF-36 questionnaire will be re-collected at 1, 2, 3, 4, and 6 months after the injection session.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 y/o or greater,
* Subacute bilateral cervical/ upper back pain, pain of longer than 2 months and shorter than 6 months duration,
* VAS pain score of 5 or greater for the cervical/ upper back pain for 4 week period before injection,
* If female or child bearing potential, concurrent use of a reliable method of contraception.

Exclusion Criteria:

* Known allergy or sensitivity to Botulinum toxin type A.
* Any medical condition that may put the subject at increased risk with exposure to BOTOX®, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
* Use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function
* Pregnancy, breast feeding, or planned pregnancy
* Acute or operative pathology on cervical MRI
* History of treatment for gatro-esophageal reflux disease
* Abnormal finding on 3-oz water swallowing test on the initial screening visit

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2006-07

PRIMARY OUTCOMES:
NDI, VAS, SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Date, MD, Principal Investigator — VA Palo Alto Health Care System; Henry Lew, MD, Ph.D, Principal Investigator — VA Palo Alto Health Care System